CLINICAL TRIAL: NCT05913570
Title: Cadonilimab as Neoadjuvant Therapy in Resectable Stage II-III Mismatch Repair-deficient (dMMR)/ Microsatellite Instability-high (MSI-H) Colorectal Cancer
Brief Title: Cadonilimab as Neoadjuvant Therapy in Resectable Stage II-III MSI-H/dMMR Colorectal Cancer
Acronym: MSI-H/dMMR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LiuYing (Other Government)
Responsible Party: Sponsor-Investigator, LiuYing, Clinical Professor, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-061-002
Record Dates: First submitted 2023-06-06; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Mismatch Repair-deficient (dMMR); Microsatellite Instability-high (MSI-H); Neoadjuvant Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Turcot syndrome | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Masking Description: Cadonilimab was approved in China in June 2022 for use in patients with relapsed or metastatic cervical cancer (r/mCC) who have progressed on or after platinum-based chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Cadonilimab (®), a PD-1/CTLA-4 bi-specific antibody (Experimental): Neoadjuvant therapy with Cadonilimab
  Interventions: Drug: Cadonilimab (®), a PD-1/CTLA-4 bi-specific antibody

INTERVENTIONS:
Drug: Cadonilimab (®), a PD-1/CTLA-4 bi-specific antibody — 10mg/kg, Q3W for 4 cycles
  Other Names: Neoadjuvant therapy with Cadonilimab

SUMMARY:
This study will evaluate the safety, and tolerability of Cadonilimab as neoadjuvant treatment for resectable local advanced colorectal cancer patient with dMMR/MSI-H.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common malignant tumours of human beings. Mismatch Repair-deficient (dMMR)/ Microsatellite Instability-high (MSI-H) CRC is a specific subtype of CRC, which accounts for approximately 15% ~20% of all CRC patients,and can not benefit from 5-fluorouracil (5-FU) adjuvant chemotherapy. Once patients have distant metastases, they are not sensitive to traditional palliative chemotherapy, and thus lead to much worse prognosis than that of mismatch repair-proficient (pMMR)/ microsatellite stability (MSS). Neoadjuvant immunotherapy based on mismatch repair (MMR) status in CRC have reported some encouraging data. The NICHE study showed that 20 CRC patients with dMMR achived pathological remission, of which 19 patients with residual tumor ≤10%, 15 patients achived pathological complete remission. Another study (ClinicalTrials.gov, NCT03926338) which investigating the effect of neoadjuvant PD-1 blockade with toripalimab, with or without celecoxib, on mismatch repair-deficient or microsatellite instability-high, locally advanced, colorectal cancer. The result revealed that all 34 patients had an R0 resection. 15 of 17 patients (88%) in the toripalimab plus celecoxib group and 11 of 17 patients (65%) in the toripalimab monotherapy group had a pathological complete response.

Cadonilimab (®), a PD-1/CTLA-4 bi-specific antibody, is being developed by Akeso, Inc. for the treatment of a range of solid tumours, including cervical cancer, lung cancer, gastric/gastroesophageal junction cancer, oesophageal squamous cell cancer, liver cancer and nasopharyngeal cancer. Cadonilimab was approved in China in June 2022 for use in patients with relapsed or metastatic cervical cancer (r/mCC) who have progressed on or after platinum-based chemotherapy.

Given the reported efficacy data about immunotherapy as neoadjuvant treatment in MSI-H/dMMR CRC, the aim of this study was to investigate the efficacy and safety of Cadonilimab as neoadjuvant treatment for resectable local advanced colorectal cancer patient with the dMMR/MSI-H.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Male or female subjects > 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histological or cytological documentation of adenocarcinoma of the colon or rectum; Tumor tissues were identified as mismatch repair-deficient (dMMR) by immunohistochemistry (IHC) method or microsatellite instability-high (MSI-H) by polymerase chain reaction (PCR) in local site; For colon cancer must be determined by CT or MRI scans as locally advanced (T4) or cN1-2 [with the definition of a clinically positive lymph node being any node ≥ 1.0 cm]). Participants should be eligible for radical resection of R0.
5. At least one measurable lesion as defined by RECIST 1.1
6. Willing and able to provide 2ml blood and archived tumor tissue sample for MSI status testing. Patients who do not have adequate archival tumor tissue available should undergo a fresh tumor biopsy
7. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment.
8. Willingness of men and women of reproductive potential to observe conventional and effective birth control for the duration of treatment and for 120 days following the last dose of study treatment; this may include barrier methods such as condom or diaphragm with spermicidal gel.

Exclusion Criteria:

1. Previous any systemic anticancer therapy for colorectal cancer disease, including chemotherapy, radiothapy or immunotherapy
2. Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody, anti-cytotoxic T lymphocyte-associated antigen 4 (cytotoxic T-lymphocyte-associated Protein 4, CTLA-4) antibody or other drug/antibody that acts on T cell costimulation or checkpoint pathways.
3. Subjects with known allergy to monoclonal antibodies
4. Previous or concurrent cancer that is distinct in primary site or histology from colon cancer within 2 years prior to study drug treatment.
5. Concurrent with active autoimmune disease or Participants with a history of autoimmune disease who may recur
6. Subjects receiving immunosuppressive agents (such as steroids, or corticosteroids at physiologic replacement doses, equivalent to ≤ 10 mg prednisone daily ) for any reason within 14 days before the study drug treatment.
7. Uncontrolled hypertension or hyperglycemia within 14 days before the study drug treatment.
8. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrent within 14 days of study drug treatment)
9. History of interstitial lung disease, noninfectious pneumonia, or poorly controlled lung disease (including pulmonary fibrosis, acute lung disease).
10. Active systemic bacterial, viral, or fungal infection， requiring systemic treatment within 14 days before study drug treatment.
11. Positive test for hepatitis B virus surface antigen with HBV DNA> 500 IU/mL（> 2500copies/mL）at screening or untreated Chronic hepatitis B
12. Positive test for hepatitis C virus ribonucleic acid (if antihepatitis C virus antibody tested positive) at screening;
13. Known history of testing positive for human immunodeficiency virus (HIV)
14. Major surgery for any reason, except diagnostic biopsy, within 28 days of the first administration of study drug. The subject must fully recovered from prior treatment before the first administration of study drug
15. Previous allogeneic stem cell transplantation or organ transplantation
16. Previous history of myocarditis, cardiomyopathy, and malignant arrhythmias
17. Vaccination within 4 weeks of the first administration of study drug and throughout the study is prohibited, except for administration of inactivated vaccines (eg, inactivated influenza vaccines).
18. All other underlying medical condition (including laboratory abnormalities) that is detrimental to study drug administration, or may affect drug toxicity or AE interpretation, or may result in inadequate or reduced adherence to study drug; Alcohol or drug abuse or dependence
19. Pregnancy or lactation
20. Concurrent participated in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rates | 1 year
  Proportion of patients experiencing a pCR to perioperative PD-1/CTLA-4 bi-specific antibody

SECONDARY OUTCOMES:
Major pathological response rates | 1 year
  The proportion of patients experiencing a major pathological response to perioperative PD-1/CTLA-4 bi-specific antibody
R0 resection rates | 1 year
  The proportion of patients experiencing a R0 resection after perioperative treatment with PD-1/CTLA-4 bi-specific antibody
Relapse-free survival (DFS) | 3 years
  Defined as the time from radical surgery to relapse, metastasis or death from any cause
The incidence of Treatment-related Adverse Events | 1 year
  Assessed by evaluation of treatment-related adverse events
Number of participants with any treatment-related delays in the planned surgery of no more than 28 days after the last preoperative Cadonilimab dose | 1 year
  Any treatment-related delays in the planned surgery of no more than 28 days after the last preoperative Cadonilimab dose

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, MD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No